CLINICAL TRIAL: NCT06299189
Title: A Therapist Guided Internet-delivered Treatment for Adults With ADHD - an Open Effectiveness Trial in Routine Care
Brief Title: A Therapist Guided Internet-delivered Treatment for Adults With ADHD (Attention Deficit / Hyperactivity Disorder) - an Open Effectiveness Trial in Routine Care
Acronym: MinADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 309264
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: ADHD; ADHD - Combined Type; ADHD Predominantly Inattentive Type; ADHD, Predominantly Hyperactive - Impulsive
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A self-guided internet delivered intervention (Experimental): MinADHD: 7 self-help modules Interventions: Behavioural
  Interventions: Behavioral: MinADHD

INTERVENTIONS:
Behavioral: MinADHD — Guided self-help, 7 modules Interventions

SUMMARY:
The primary objective of this study is to explore and evaluate the use and utility of a guided Internet-delivered psychological treatment for adults with ADHD with a combined focus on:

i) Evaluating the impact of potential predictors to treatment adherence, treatment response, treatment use and utilty. ii) Evaluating the feasibility, clinical benefits and implementation process of the treatment in routine outpatient care. iii) Evaluate the cost-effectiveness of the treatment program.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder characterized by symptoms of inattention and/or hyperactivity/impulsivity that are persistent across time and situations. ADHD in adulthood, with estimated prevalence of 2-3%, is associated with challenges that may have severe consequences on daily life functioning. Treatments delivered over the Internet on smartphones or personal computers may help to increase the availability of effective psychological interventions for a larger group of adults with ADHD. The overall aim of this study is to investigate 1) predictors of effect; 2) implementation outcomes; and the 3) cost-benefit of a therapist guided Internet-delivered treatment for adults with an ADHD diagnosis. The study is an open longitudinal cohort trial in routine care. A total of 200 participants with an ADHD diagnosis will be included in the trial, and 15 participants will be interviewed about their experiences with guided Internet-delivered treatment. The outcomes are change in primary and secondary symptoms and quality of life, cost-benefit and implementation outcomes of guided internet-delivered treatment for adults with ADHD. The investigators will use quantitative statistical procedures and qualitative methods to analyze the data. The results from the study will contribute to the growing research on Internet-delivered treatments. The expected results may have a major impact on treatment provision and the further development of treatment options for adults with ADHD. Moreover, investigating ways to increase adoption, adherence and fidelity in Internet-delivered treatment could be of great value when implementing such treatment into routine care.

ELIGIBILITY:
Inclusion criteria: |

* Age ≥18
* A self-reported diagnosis of ADHD
* Access to and ability to use a computer, smartphone and the Internet.
* Speaks, writes and reads Norwegian

Exclusion criteria:

* In need of other psychological treatment for mental health illness such as borderline or personality disorder, bipolar disorder, substance abuse or psychosis.
* Ongoing psychological treatment for ADHD or other psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The Adult ADHD Self-Rating Scale | From enrollment to the end of 6-months follow-up
  Measure of ADHD symptom severity
Adult ADHD Quality of Life Measure | From enrollment til the end of 6-month follow-up.
  Measure of impact of ADHD on quality of life

SECONDARY OUTCOMES:
The Patient Health Questionnaire | From enrollment til the end of 6-month follow-up.
  Measure of depression
Generalized Anxiety Disorder-7 | From enrollment til the end of 6-month follow-up.
  Measure of anxiety
Personality Disorder Severity ICD-11 | From enrollment til the end of 6-month follow-up.
  Measure of personality functioning
EuroQoL 5D-5L | From enrollment to end of 6-month follow-up.
  Measure of health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Bjørgvin DPS, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
The IPD collected for the current trial is considered sensitive patient information.